CLINICAL TRIAL: NCT04988958
Title: Radical Versus Conservative Surgical Treatment of Liver Hydatid Cysts: A Propensity Score Matching Analysis
Brief Title: Radical Versus Conservative Surgical Treatment of Liver Hydatid Cysts
Status: Completed | Type: Observational
Sponsor: Université de Sousse (Other)
Responsible Party: Principal Investigator, ammar houssem, clinical professor, Université de Sousse
Other Study IDs: U23477
Record Dates: First submitted 2021-07-13; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Hydatid Cyst
MeSH Terms: conditions — Echinococcosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: hydatid cyst resection — radical resection of hydatic cyst

SUMMARY:
The management of liver hydatid cysts (LHC) is controversial. Surgery remains the basic treatment, and can be divided into radical and conservative approaches. The purpose of this study was to compare the outcome of radical and conservative surgery (CS) in the treatment of LHC and to evaluate the efficiency and safety of radical surgery (RS).

DETAILED DESCRIPTION:
The management of liver hydatid cysts (LHC) is controversial. Surgery remains the basic treatment, and can be divided into radical and conservative approaches. The purpose of this study was to compare the outcome of radical and conservative surgery (CS) in the treatment of LHC and to evaluate the efficiency and safety of radical surgery (RS).

Data from all patients with LHC treated in Sahloul Hospital, between January 2000 and December 2019, were retrieved from a retrospective database. To minimize selection bias, propensity score matching (PSM) was performed, based on variables representing patient characteristics and operative risk factors.

RS especially total pericystectomy had fewer postoperative complications and lower recurrence rate compared to CS. RS may be the preferred procedure for LHC if the expertise is available.

ELIGIBILITY:
Inclusion Criteria:

* age over 14 years old.
* Patients presenting liver hydatid cyst .

Exclusion Criteria:

* age less than 14 years old.
* Patients presenting other localization of hydtic cyst , than the liver.
* calcified cysts.
* patients with incomplete medical records.
* patients who were lost to follow up.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 914 Patients , who underwent surgical treatment at the Department of General and Digestive Surgery, Sahloul University Hospital Center, Sousse, Tunisia from 1st January 2000 to 31st December 2019 was performed. The diagnosis of LHC was established by clinical history, physical examination and abdominal ultrasonography (USG) in all patients
Sampling Method: Non-Probability Sample
Enrollment: 914 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
recurrence of hydatic cyst | 2 years
  recurrence of hydatid cyst after surgery

IPD SHARING:
Plan to Share IPD: Undecided